CLINICAL TRIAL: NCT00954135
Title: Letrozole Plus Oral Cyclophosphamide Plus/Minus Sorafenib as Primary Systemic Treatment in Post-menopausal, Estrogen Receptor Positive, Breast Cancer Patients
Brief Title: Letrozole Plus Oral Cyclophosphamide Plus/Minus Sorafenib as Primary Systemic Treatment in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Alfredo Berruti, Dipartimento di Scienze Cliniche e Biologiche Università di Torino
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-006208-39
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: neoadjuvant therapy, sorafenib, letrozolo, cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozolo+cyclophosphamide (Active Comparator)
  Interventions: Drug: letrozolo+cyclophosphamide
- letrozolo+sorafenib+cyclophosphamide (Experimental)
  Interventions: Drug: letrozolo+sorafenib+cyclophosphamide

INTERVENTIONS:
Drug: letrozolo+cyclophosphamide — Letrozole 2,5 mg/daily + metronomic cyclophosphamide 50 mg/daily for 6 months
  Arms: letrozolo+cyclophosphamide
Drug: letrozolo+sorafenib+cyclophosphamide — Letrozole (2,5 mg/daily) + "metronomic" cyclophosphamide (50 mg/daily) + Sorafenib (400 mg/bid/daily) for 6 months
  Arms: letrozolo+sorafenib+cyclophosphamide

SUMMARY:
Endocrine therapy is the mainstay of systemic treatment in patients with endocrine responsive breast cancer. Aromatase inhibitors are the most active agents in post-menopausal women. Randomized comparisons either in primary/adjuvant setting or in metastatic disease setting have demonstrated the superiority of these drugs over tamoxifen.

Primary systemic treatment administered to breast cancer patients is a useful model to identify baseline features able to predict which patients are most likely to benefit from cytotoxic treatment and is a way to study new biological markers in relation to the predictive information they provide.

This treatment modality represents therefore the best way to explore new treatment strategies in particular treatment strategies involving target therapies.

We have conducted a randomised phase II trial in which the activity of Letrozole plus/minus oral metronomic cyclophosphamide as primary systemic treatment has been investigated in a patient population of elderly breast cancer patients. The conclusions were that the combination of letrozole with metronomic cyclophosphamide was a very active scheme. In addition this was the first study demonstrating in vivo the antiangiogenic effect of metronomic scheduling. This study suggests that chemotherapy administered on a metronomic schedule, targeting therefore the neo-angiogenesis, could be synergistic with endocrine therapy with aromatase inhibitors.

Sorafenib is a multi-kinase inhibitor targeting Raf, VEGFR-1, VEGFR-2, VEGFR-3, PDGFR-alfa, Flt-3, c-Kit, and p38.

There is a strong rationale of combining different anti-angiogenic agents. At the ASCO 2007 meeting the data of a phase I study exploring the toxicity of a combination of sorafenib and bevacizumab have been presented. The results showed an increased toxicity being dose limiting in some patients. To our knowledge there are no data un activity and toxicity of adding sorafenib to metronomic chemotherapy.

DETAILED DESCRIPTION:
Primary Objective:

To compare the activity of the 2 regimens The primary end point will be the clinical complete response rate of each treatment arm among all registered cases (intent to treat analysis).

Secondary Objectives:

To compare the 2 treatment arms with respect to:

* Toxicity
* Progression Free Survival
* Overall survival

Ancillary studies To evaluate before and after treatment a number of markers of hypoxia, neoangiogenesis, apoptosis, EGFR activating pathways.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women in postmenopausal status
* 2. Age> 60 or age > 18 and unfit for chemotherapy with commonly employed regimens in breast cancer patients
* 3. Diagnosis of invasive BC, T>2, N0-N2, M0,
* 4. Endocrine Responsive disease according to San Gallen criteria
* 5. ECOG Performance Status of 0 or 2
* 6. Life expectancy of at least 12 weeks
* 7. In case of recent surgery, the wound must be completely healed prior to receiving Sorafenib
* 8. Subjects with at least one uni-dimensional(for RECIST) or bi-dimensional(for WHO) measurable lesion. Lesions must be measured by CT-scan or MRI
* 9. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* 10. Hemoglobin > 9.0 g/dl
* 11. Absolute neutrophil count (ANC) >1,500/mm3
* 12. Platelet count 100,000/μl
* 13. Total bilirubin < 1.5 times the upper limit of normal
* 14. ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
* 15. Alkaline phosphatase < 4 x ULN
* 16. PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
* 17. Serum creatinine < 1.5 x upper limit of normal.

Exclusion Criteria:

* 1. History of cardiac disease:congestive heart failure >NYHA class 2;active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy( beta blockers or digoxin are permitted) or uncontrolled hypertension.
* 2. History of HIV infection or chronic hepatitis B or C (This criteria should be modified to allow Hepatitis B or C in protocols looking at HCC patient population).
* 3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* 4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* 5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* 6. History of organ allograft The organ allograft may be allowed as protocol specific.
* 7. Patients with evidence or history of bleeding diathesis
* 8. Patients undergoing renal dialysis
* 9. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | six years

SECONDARY OUTCOMES:
Overall survival | six years

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, MD, Study Chair — Medical Oncology, Department of clinical and biological sciences Univerity of Turin; Daniele Generali, MD, Principal Investigator — Breast Unit Azienda Ospedaliera Istituti Ospitalieri Cremona; Alberto Bottini, MD, Study Director — Breast Unit Azienda Ospedaliera Istituti Ospitalieri Cremona
Locations (2):
- Italy (2):
  - Breast Unit Azienda Ospedaliera Istituti Ospitalieri, Cremona
  - Azienda Ospedaliera S.Luigi Orbassano, Orbassano

REFERENCES:
- [Result] Bottini A, Generali D, Brizzi MP, Fox SB, Bersiga A, Bonardi S, Allevi G, Aguggini S, Bodini G, Milani M, Dionisio R, Bernardi C, Montruccoli A, Bruzzi P, Harris AL, Dogliotti L, Berruti A. Randomized phase II trial of letrozole and letrozole plus low-dose metronomic oral cyclophosphamide as primary systemic treatment in elderly breast cancer patients. J Clin Oncol. 2006 Aug 1;24(22):3623-8. doi: 10.1200/JCO.2005.04.5773. PMID 16877730